CLINICAL TRIAL: NCT05121337
Title: Effects of DASH Groceries on Blood Pressure in Black Residents of Urban Food Deserts Without Treated Hypertension
Brief Title: Groceries for Black Residents of Boston to Stop Hypertension Among Adults Without Treated Hypertension
Acronym: GoFresh
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Stephen Juraschek, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021P000825; GEMS # 42359 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2021-10-25; First posted 2021-11-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Elevated Blood Pressure; Hypertension
Keywords: hypertension; blood pressure; nutrition; diet; DASH; sodium; trial; dietitian; cholesterol
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Individual level, parallel, randomized trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcomes assessors will not know randomization assignment. Investigators will not know randomization assignment. Participants and the nutritionist/dietitian interventionist will need to know randomization assignment in order to carry out the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietitian-Assisted DASH groceries (Experimental): Participants will order groceries sufficient to meet their caloric needs each week for 12 weeks with the assistance of a dietitian/nutrition interventionist. Groceries will be delivered to participants' homes or picked up at a convenient location. The dietitian/nutrition interventionist will provide brief educational content at the time of food delivery. Orders will be placed via phone or through virtual counseling sessions. During the remainder of the study (months 4-12), participants will be asked to apply what they learned without the provision of groceries.
  Interventions: Behavioral: Dietitian-Assisted DASH groceries
- Self-directed shopping (referent assignment) (Active Comparator): Participants will receive a monthly stipend over a 3 month period and some basic information about healthy eating. The stipend is not restricted to foods. During the remainder of the study (months 4-12), participants will be asked to continue their typical shopping without the provision of the monthly stipend.
  Interventions: Behavioral: Self-directed shopping

INTERVENTIONS:
Behavioral: Dietitian-Assisted DASH groceries — The DASH ("Dietary Approaches to Stop Hypertension"), is a healthy dietary pattern that lowers blood pressure without reducing weight. The DASH diet emphasizes fruits, vegetables, and low-fat dairy products; includes whole grains, poultry, fish, and nuts; and is reduced in red meat, sweets, and sugar-containing beverages.
  Intervention Phase:
  This intervention is a weekly, 12-week DASH dietary intervention. A dietitian will assist participants in ordering groceries in a pattern consistent with the DASH diet to be delivered to their homes. The quantity of groceries will be based on participant Calorie needs and family size.
  Observation Phase:
  For months 4-12 of the study, participants will be asked to continue following a DASH grocery shopping pattern without the provision of weekly groceries.
  Arms: Dietitian-Assisted DASH groceries
Behavioral: Self-directed shopping — Intervention Phase:
  Participants will receive some basic information on healthy eating and a monthly stipend at 4, 8, and 12-weeks of the intervention.
  Observation Phase:
  For months 4-12 of the study, participants will be asked to follow their typical shopping pattern without the provision of a monthly stipend.
  Arms: Self-directed shopping (referent assignment)

SUMMARY:
GoFresh is a randomized trial, testing the effects of a home-delivered DASH-patterned grocery intervention on blood pressure in Black adults, residing in Boston area urban food deserts.

DETAILED DESCRIPTION:
Hypertension affects over half of Black adults in the United States - more than any other group - and diet is a principal determinant of disparities in hypertension among Black adults. While the DASH diet is a proven strategy for lowering blood pressure in Black adults, diet disparities are increasing in urban food deserts due to poor access and the high costs of healthy foods. This clinical trial will randomize 150 Black adults residing in Boston area urban food deserts to either:

1. 12 weeks of dietitian-assisted, DASH grocery delivery via an online, virtual grocery store at an amount sufficient to replace all Calorie needs of each participant, allowing for some sharing with family members

   or
2. Self-directed shopping with a monthly stipend over a 3-month period

After the 12-week intervention phase, participants will undergo a 9-month observation phase. At 3-months after the intervention is complete the investigators will repeat in-person study assessments and perform qualitative interviews in a subset of the population to determine barriers and facilitators to intermediate-term maintenance of the intervention. At 9-months after the intervention, participants will participate in a phone visit designed to assess longer-term maintenance of the intervention.

ELIGIBILITY:
INCLUSION:

* Self-reported/self-identified as Black or African American
* Resting systolic blood pressure of 120 to <150 mm Hg and diastolic blood pressure <100 mm Hg
* Residence in communities identified as Boston area food deserts: Brighton, Chelsea, Dorchester, East Boston, Everett, Hyde Park, Jamaica Plain, Malden, Mattapan, Revere, Roslindale, Roxbury, or Winthrop
* Able to receive home-delivered groceries or pick them up at a convenient location and willing to eat only the groceries provided over a 12-week period
* Have access to refrigeration, cooking appliances, and Wi-Fi/cellular service
* Have access to mobile device or computer to be able to conduct grocery orders via video conference or by phone
* Willing and able to complete required measurement procedures

EXCLUSION:

Laboratory Exclusions:

* Serum potassium ≥5.0 mmol/L or <3.5 mmol/L
* Estimated glomerular filtration rate (eGFR) <30 mL/min per 1.73 m^2 by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
* Hemoglobin A1c ≥6.5%

Medication Exclusions:

* Any use of medications that lower blood pressure or medications intended for hypertension treatment (including antihypertensives taken for non-hypertension purposes) within the last 6 months
* Unstable doses (i.e. a change in the 2 months prior to screening or randomization) of the following:

  * Sodium-glucose co-transporter 2 (SGLT2) inhibitors
  * Stimulants
  * Inhaled or oral medications for asthma or chronic obstructive pulmonary disease (COPD)
  * Hormone replacement therapy or thyroid hormone
  * Weight-increasing psychotropic agents, including antipsychotic agents, lithium, and mirtazapine
* Use of any of the following medications:

  * Potassium supplement, except if part of a multivitamin
  * Warfarin (Coumadin)
  * Chronic oral corticosteroid (intermittent use is okay)
  * Weight loss medications (including GLP-1 receptor agonists)
* Unwillingness to keep same dose of vitamin, mineral, and botanical supplements
* Any medication not compatible with participation as determined by the investigators

Physical Exclusions:

* Systolic blood pressure ≥150 mm Hg or diastolic blood pressure ≥100 mm Hg
* Body weight >420 pounds
* Arm circumference >50cm
* Weight loss or gain of >5.0% of body weight during prior 2 months

Medical History Exclusions:

* Type 1 or Type 2 Diabetes defined as a hemoglobin A1c ≥6.5% or diabetes treatment
* Active cardiovascular disease or any event in the prior 6 months, including coronary artery bypass grafting (CABG), percutaneous transluminal coronary angioplasty (PTCA), myocardial infarction (MI), cerebrovascular accident (CVA), or congestive heart failure (CHF) exacerbation requiring hospital admission
* Cancer diagnosis or treatment in the last 2 years (non-melanoma skin cancer or localized breast or prostate or bladder cancer not requiring systemic therapy is acceptable)
* Active inflammatory bowel disease, bowel resection, malabsorptive syndrome, pancreatitis (episode within past year), or history of bariatric surgery
* Pregnancy or lactation or planned pregnancy
* Any emergency department (ED) visit for asthma or chronic obstructive pulmonary disease (COPD) in the last 6 months
* Any other serious illness or condition not compatible with participation as determined by the investigators

Lifestyle and Other Exclusions:

* Significant food allergies, preferences, intolerances, or dietary requirements that would interfere with diet adherence
* Consumption of more than 14 alcoholic drinks per week or consumption of more than 6 drinks on one or more occasion per week
* Active substance use disorder that would interfere with participation
* Extreme food insecurity
* Participation in or planning to start weight loss program
* Current participation in another clinical trial that could interfere with the study protocol
* Anticipated change in residence prior to the end of the study
* Families with more than 6 adults at dinner time (children are considered to be half an adult)
* Investigator discretion

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Seated, office-based, systolic blood pressure (intervention phase) | Measured 3 months after randomization
  In-person, measured with an automated oscillometric device that will perform 3 measurements.

SECONDARY OUTCOMES:
Seated, office-based, systolic blood pressure (observation phase) | Measured 6 months after randomization
  In-person, measured with an automated oscillometric device that will perform 3 measurements.
Seated, office-based, diastolic blood pressure (intervention & observation phases) | Measured 3 and 6 months after randomization
  In-person, measured with an automated oscillometric device that will perform 3 measurements.
Ambulatory blood pressure monitoring: wake-time systolic and diastolic blood pressure (intervention & observation phases) | Measured 3 and 6 months after randomization
  Ambulatory blood pressure monitoring with a mobile blood pressure device that will measure blood pressure over a 24-hour period.
Body Mass Index (BMI) (intervention & observation phases) | Measured 3 and 6 months after randomization
  In-person, measurement based on height and weight. Height is measured via a stadiometer and weight is measured via calibrated scale.
24-hour urine potassium (intervention & observation phases) | Measured 3 and 6 months after randomization
  Collected at home after a clinic void over a 24-hour period
24-hour urine sodium (intervention & observation phases) | Measured 3 and 6 months after randomization
  Collected at home after a clinic void over a 24-hour period
Hemoglobin A1c (intervention & observation phases) | Measured 3 and 6 months after randomization
  In-person blood collection; measure of glycemia over the preceding 3 months
Lipids (intervention & observation phases) | Measured 3 and 6 months after randomization
  Measured in fasted serum specimens collected during phlebotomy. Includes total cholesterol, high density lipoprotein cholesterol, derived low density lipoprotein cholesterol, and triglycerides
Serum potassium (intervention & observation phases) | Measured 3 and 6 months after randomization
  Measured in blood as part of a basic metabolic panel
Serum creatinine (intervention & observation phases) | Measured 3 and 6 months after randomization
  Measured in blood as part of a basic metabolic panel
Daily intake of fat, fruits, and vegetables (intervention & observation phases) | Measured 3, 6, and 12 months after randomization
  Assessed via questionnaire in-person and via phone call; assessed via a validated food screener (Block et al; PMID: 10788730).
24-hour dietary recall (intervention & observation phases) | Measured 3 and 6 months after randomization
  Assessed via questionnaire in-person using the Automated Self-Administered 24-Hour Dietary Recall (ASA24)

OTHER OUTCOMES:
Qualitative Interviews | 6 months after randomization
  The investigators will perform qualitative interviews in a subpopulation of both study assignments to assess for barriers and facilitators related to long-term maintenance of the intervention.
Short Form 12 Item Health Survey (SF-12) | Measured 3, 6, and 12 months after randomization
  Assessment of global health-related quality of life
Grocery shopping and dining habits | Measured 3, 6, and 12 months after randomization
  This is a modified version of the interviewer-administered SHoPPER (Study of Household Purchasing Patterns, Eating, and Recreation) instrument (French et al; PMID: 30808311) with some modifications to assess grocery shopping, meal preparation, and dining behaviors and habits.
Perceived Stress Scale 4 (PSS-4) | Measured 3, 6, and 12 months after randomization
  An instrument used to assess participants' feelings about stress

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Juraschek, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center - Clinical Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
This project is one of five projects that form the AHA's AddREssing Social Determinants TO PRevent HypErtension (RESTORE) Network. A de-identified database will be provided for use by investigators external to BIDMC upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6-12 months after the study is complete
Access Criteria: Upon reasonable request to investigators.

REFERENCES:
- [Background] Turkson-Ocran RN, Cluett JL, Fitzpatrick SL, Kraemer KM, McManus K, Mukamal KJ, Davis RB, Elborki M, Ferro K, Ismail N, Laura Aidoo E, Larbi Kwapong F, Castilla-Ojo N, Grobman B, Seager R, Hines AL, Miller ER, Crews DC, Juraschek SP. Rationale and Design of the Groceries for Black Residents of Boston to Stop Hypertension Among Adults Without Treated Hypertension (GoFresh) Trial. Am J Hypertens. 2023 Apr 15;36(5):256-263. doi: 10.1093/ajh/hpad008. PMID 37061794
- [Derived] Ferro KM, Seager R, McManus K, Kraemer KM, Turkson-Ocran RAN, Michetti J, Allison S, Fitzpatrick S, Juraschek SP. Nutrition intervention of groceries for Black residents of Boston to stop hypertension (GoFresh) among adults with or without treated hypertension trial: rationale, design, and guiding domains. Trials. 2025 Dec 3;26(1):560. doi: 10.1186/s13063-025-09273-z. PMID 41340057
- [Derived] Juraschek SP, Col H, Ferro K, Turkson-Ocran RN, Cluett JL, Davis RB, Kraemer KM, McManus K, Mukamal KJ, Aidoo EL, Larbi Kwapong F, Budu M, Patil D, Nartey S, Michetti J, Allison S, Mate-Kole M, Cao J, Grobman B, Seager R, Hines AL, Miller ER 3rd, Crews DC, Fitzpatrick SL; GoFresh Collaborative Research Group. DASH-Patterned Groceries and Effects on Blood Pressure: The GoFresh Randomized Clinical Trial. JAMA. 2026 Jan 6;335(1):36-48. doi: 10.1001/jama.2025.21112. PMID 41206973
- [Derived] Harry T, Hussain Z, Cao J, Turkson-Ocran RN, Juraschek SP, Michos ED, Miller HN, Lahey TP, Plante TB, Feng Y. Randomized Comparison of Online Motivational Themes in Clinical Trial Recruitment. Circ Cardiovasc Qual Outcomes. 2025 Dec;18(12):e012945. doi: 10.1161/CIRCOUTCOMES.125.012945. Epub 2025 Nov 7. PMID 41201904
- See also: Main trial website — http://gofreshstudy.org

DOCUMENTS (2):
  • Study Protocol (2025-03-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT05121337/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT05121337/SAP_001.pdf